CLINICAL TRIAL: NCT04317495
Title: Augmenting Repetitive Transcranial Magnetic Stimulation (rTMS) With Cognitive Control Training in Major Depressive Disorder (MDD)
Brief Title: Augmenting rTMS With Cognitive Control Training in Major Depressive Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: New data has caused the principal investigator to decide that the study no longer makes sense to conduct as it is designed. This is not a suspension of IRB approval.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Stephan F. Taylor, Professor of Psychiatry, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00161598
Record Dates: First submitted 2020-03-19; First posted 2020-03-23 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Major Depressive Disorder
Keywords: transcranial magnetic stimulation; computerized cognitive training
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Computerized Cognitive Training (CCT) (Experimental): The patients will receive CCT during their standard rTMS treatments (after having 5 days of treatment until the pre-taper treatment).
  Interventions: Other: Computerized Cognitive Training (CCT)

INTERVENTIONS:
Other: Computerized Cognitive Training (CCT) — After having four rTMS sessions without CCT, the patients will perform CCT (starting day 5) during the rTMS session, which typically last from 20-40 minutes. A course of rTMS therapy includes from 25-36 treatments, given daily, until the last 5-6 treatments, given as a 'taper' over 2 weeks. CCT will be paired with rTMS up until the taper begins. In addition, they will have assessments prior to and after the therapy.

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) is an effective treatment for MDD, but the overall effect sized of the treatment is equivalent to antidepressant pharmacotherapy, and responses are highly variable. Given that rTMS is usually given to patients who have failed pharmacotherapy, a more effective alternative is needed.

Therefore, this study will combine computerized cognitive training (CCT) during standard rTMS treatments and assess its feasibility, tolerability, and changes in cognitive control performance and depression symptoms.

Participants that agree to the study and meet eligibility will receive standard rTMS (generally 25-36 daily treatments) along with CCT (starting on day 5 of treatment until the pre-taper treatment). In addition, to CCT participants will be asked to complete assessments before and after treatment

DETAILED DESCRIPTION:
This project will also have a registry for participants that are approached to be in the clinical trial with the CCT but don't wish to be enrolled. Although the registry will be available for these participants, the information entered into this ClinicalTrials.gov registration will reflect the clinical trial portion of this project.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder
* Eligible to receive and recommended for rTMS for depression
* Willingness to complete computerized cognitive training and undergo brain stimulation procedures
* Must be enrolled as a Michigan Medicine patient and currently receiving TMS treatment as part of your clinical care.

Exclusion Criteria:

* History of serious neurological illness or brain injury (e.g., stroke)
* Poor visual acuity impairing performance on the computerized tasks (eyeglasses must be removed for rTMS treatment, but contacts are permissible)
* Diagnosed intellectual disability
* Inability to manipulate a tablet device while seated in the rTMS chair

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Feasibility assessed by percentage of CCT sessions completed during rTMS | approximately 30 days (usually 20-30 sessions)
  Percentage CCT sessions completed: (number of sessions completed/number of sessions assigned) X 100

SECONDARY OUTCOMES:
Time on task during treatment | For each day: 45 min; for entire treatment: approx 30 days
  Percentage time on task: (Time engaged with task/total time of task assigned)X100, averaged over all active sessions
Acceptability of CCT | through study completion date, up to 2 years
  Percentage: (Number of eligible patients accepting CCT/number of patients approached but not accepting CCT) x 100
Cognitive Control Performance change over course of treatment | Approximately 30 days (usually 20-30 sessions)
  Average percentage correct trials on n-back working memory task for first 2 sessions minus average percentage correct trials for last 2 sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Taylor, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No